CLINICAL TRIAL: NCT07215832
Title: Karyopharm Expanded Access Program for Selinexor
Acronym: KEAP
Status: Available | Type: Expanded Access
Sponsor: Karyopharm Therapeutics Inc (Industry)
Collaborators: Caligor Coghlan (CalCog) (Unknown)
Responsible Party: Sponsor
Other Study IDs: KEAP-KPT-330
Record Dates: First submitted 2025-09-30; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma; Diffuse Large B-Cell Lymphoma (DLBCL); Sarcoma; Neuroglioblastoma; Peripheral T-cell Lymphoma; Endometrial Cancer; Myelofibrosis; Other
Keywords: selinexor
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Large B-Cell, Diffuse; Sarcoma; Lymphoma, T-Cell, Peripheral; Endometrial Neoplasms; Primary Myelofibrosis | interventions — selinexor

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: selinexor
  Other Names: KPT-330

SUMMARY:
KEAP is an expanded access program designed to provide selinexor to eligible participants outside of a clinical trial before the drug has been given marketing approval by the country's regulatory agency or the drug is commercially available in the country. Patients who do not qualify for an ongoing clinical trial but who might benefit from the investigational medicine may be eligible, provided they have exhausted all other available treatment options. Investigational medicines are provided to patients only through treating physicians who obtain the relevant approval on behalf of their patient from the relevant regulatory agency and follow all applicable safety-reporting regulations of the respective country.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult